CLINICAL TRIAL: NCT01249066
Title: Expression of AMP-activated Protein Kinase (AMPK) Protein in Lung Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Fang Hsin-Yuan/Director, China Medical University Hospital
Other Study IDs: DMR99-IRB-096
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-09

CONDITIONS: Lung Adenocarcinoma
Keywords: AMP-activated protein kinase; lung adenocarcinomas; Prognosis; Observation study
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
AMP-activated protein kinase (AMPK) is an evolutionally conserved protein kinase that serves as an energy guardian to help cells adapt to various metabolic stress including hypoxia. Because the role of AMPK in cancers has not been fully elucidated, in this study we investigated the expression and activation of AMPK in lung adenocarcinoma (LADC) cells and tissue.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer received operation lobectomy in CMUH

Exclusion Criteria:

* History of uremia, other malignant disease, and liver cirrhosis
* History of pneumonia and pulmonary tuberculosis
* History of long period of medications.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer received lobectomy in CMUH
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Locations (1):
- Fang Hsin Yuan, Taichung, Taiwan